CLINICAL TRIAL: NCT00880620
Title: A Placebo-Controlled Study To Evaluate The Safety And Efficacy Of IPX066 In Subjects With Parkinson's Disease
Brief Title: A Study To Evaluate The Safety And Efficacy Of IPX066 In Subjects With Parkinson's Disease
Acronym: APEX-PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPX066-B08-05
Record Dates: First submitted 2009-04-03; First posted 2009-04-14 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2017-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): One Placebo capsule was given TID for the first 21 days. Two placebo capsules were given TID on days 22 till end of study (week 30).
  Interventions: Drug: Placebo
- IPX066 145 mg LD (Experimental): One IPX066 95 mg LD was given TID on days 1-3. One IPX066 145 mg LD was given TID on days 4-21. One IPX066 145 mg LD and one placebo capsule were given TID on days 22 till end of study (week 30).
  Interventions: Drug: Placebo; Drug: IPX066 95 mg LD; Drug: IPX066 145 mg LD
- IPX066 245 mg LD (Experimental): One IPX066 95 mg LD was given TID on days 1-3. One IPX066 145 mg LD was given TID on days 4-7. One IPX066 195 mg LD was given TID on days 8-14. One IPX066 245 mg LD was given TID on days 15-21. One IPX066 245 mg LD and one placebo capsule were given TID on days 22 till end of study (week 30).
  Interventions: Drug: Placebo; Drug: IPX066 95 mg LD; Drug: IPX066 145 mg LD; Drug: IPX066 195 mg LD; Drug: IPX066 245 mg LD
- IPX066 390 mg LD (Experimental): One IPX066 95 mg LD was given TID on days 1-3. One IPX066 145 mg LD was given TID on days 4-7. One IPX066 195 mg LD was given TID on days 8-14. One IPX066 245 mg LD was given TID on days 15-21. Two IPX066 195 mg LD capsules were given TID on days 22 till end of study (week 30).
  Interventions: Drug: IPX066 95 mg LD; Drug: IPX066 145 mg LD; Drug: IPX066 195 mg LD; Drug: IPX066 245 mg LD

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: IPX066 145 mg LD; IPX066 245 mg LD; Placebo
Drug: IPX066 95 mg LD — IPX066 capsule containing 95 mg LD/23.75 mg CD
  Other Names: CD-LD ER 95 mg
  Arms: IPX066 145 mg LD; IPX066 245 mg LD; IPX066 390 mg LD
Drug: IPX066 145 mg LD — IPX066 capsule containing 145 mg LD/36.25 mg CD
  Other Names: CD-LD ER 145 mg
  Arms: IPX066 145 mg LD; IPX066 245 mg LD; IPX066 390 mg LD
Drug: IPX066 195 mg LD — IPX066 capsule containing 195 mg LD/48.75 mg CD
  Other Names: CD-LD ER 195 mg
  Arms: IPX066 245 mg LD; IPX066 390 mg LD
Drug: IPX066 245 mg LD — IPX066 capsule containing 245 mg LD/61.25 mg CD
  Other Names: CD-LD ER 245 mg
  Arms: IPX066 245 mg LD; IPX066 390 mg LD

SUMMARY:
This study examines the efficacy of three doses of IPX066 as compared to placebo in Parkinson's disease.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, fixed-dose, parallel-arm study of three doses of IPX066 versus placebo.

Total of 427 subjects were screened and 381 were randomized and received one of the four treatment groups (1) placebo (N=92), (2) IPX066 145 mg LD (N=87) (3) IPX066 245 mg LD (N=104) (4) IPX066 390 mg LD (N=98) three times a day.

Study duration is approximately 30 weeks for each subject including 4 weeks of titration (up to 3 weeks of dose escalation and I week of stabilization for safe escalation to the allocated dose), and 26 weeks of maintenance.

During the titration phase:

The following dose strengths were used to titrate up to the final three strengths that were assigned to the three IPX066 treatment arms.

IPX066 95 mg LD capsule containing 95 mg LD and 23.75 mg CD. IPX066 145 mg LD capsule containing 145 mg LD and 36.25 mg CD. IPX066 195 mg LD capsule containing 195 mg LD and 48.75 mg CD. IPX066 245 mg LD capsule containing 245 mg LD and 61.25 mg CD.

During the maintenance phase:

IPX066 145 mg LD treatment arm received 145 mg LD and 36.25 mg CD. IPX066 245 mg LD treatment arm received 245 mg LD and 61.25 mg CD. IPX066 390 mg LD treatment arm received 390 mg LD and 97.50 mg CD.

Primary efficacy outcome measure was change from baseline in the sum of UPDRS Part II and Part III scores at the end of study or last value reported if subject discontinued prematurely.

Summary of Change From Baseline to End of Study in Mean Parkinson's Disease Questionnaire-39 (PDQ-39) Score.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to voluntarily sign an informed consent form (ICF) and Health Insurance Portability and Accountability Act (HIPAA) authorization or local equivalent if applicable.
2. Diagnosed with idiopathic PD.
3. LD-naïve: defined as subjects not exposed to LD or catechol-O-methyl transferase inhibitors for more than 30 days and the exposure is not within 4 weeks prior to study enrollment.
4. If currently taking anticholinergic therapy, amantadine, or a monoamine oxidase type B (MAO-B) inhibitor, maintains a stable regimen for at least 4 weeks prior to Baseline, and agrees to maintain the stable regimen throughout study participation.
5. Agrees to use a medically acceptable method of contraception throughout the study and for 1 month after completing the study.
6. Able and willing to comply with the protocol, including availability for all scheduled clinic visits and telephone calls.

Exclusion Criteria:

1. Pregnant or breastfeeding.
2. Diagnosed with atypical Parkinsonism or any known secondary parkinsonian syndrome.
3. Prior functional neurosurgical treatment for PD or if such procedures are anticipated during study participation.
4. Use of nonselective MAO inhibitors.
5. Use of dopamine agonists within 30 days prior to Screening.
6. Unable to tolerate a placebo regimen, in the Investigator's opinion.
7. Treatment of psychosis with any antipsychotic.
8. History of seizure or epilepsy.
9. Active or prior medical condition or prior surgical procedure that would interfere with LD absorption.
10. History of narrow-angle glaucoma.
11. Subjects with a history of malignant melanoma.
12. History of myocardial infarction with residual atrial, nodal, or ventricular arrhythmias, upper gastrointestinal hemorrhage, or neuroleptic malignant syndrome.
13. Received any investigational medications during the 30 days prior to Screening.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2009-04; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Study Director — Impax Laboratories, LLC
Locations (60):
- United States (27):
  - University of Alabama at Birmingham, Dept. of Neurology, Birmingham, Alabama
  - HOPE Research Institute, LLC, Phoenix, Arizona
  - Collaborative NeuroScience Network, Inc., Garden Grove, California
  - Coastal Neurological Medical Group, La Jolla, California
  - Coordinated Clinical Research, La Jolla, California
  - The Parkinson's Institute, Sunnyvale, California
  - Yale Neurology Clinics, Temple Medical Center, New Haven, Connecticut
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Sunrise Clinical Research, Inc., Hollywood, Florida
  - Renstar Medical Research, Ocala, Florida
  - Charlotte Neurological Services, Port Charlotte, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - Idaho Elks Rehabilitation Hospital, Boise, Idaho
  - Rush University Medical Center, Dept. of Neurological Sciences, Chicago, Illinois
  - Landon Center on Aging, Dept. of Neurology, Parkinson's Disease Center, Kansas City, Kansas
  - Boston University School of Medicine, Boston, Massachusetts
  - Quest Research Institute, Bingham Farms, Michigan
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - UMDNJ Robert Wood Johnson Medical Center, Department of Neurology, New Brunswick, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University, New York, New York
  - State University of New York Upstate Medical University, Dept. of Neurology, Syracuse, New York
  - Duke University Medical Center Movement Disorders Center, Durham, North Carolina
  - University of Toledo, Toledo, Ohio
  - Baylor College of Medicine, Parkinson's Disease Center, Houston, Texas
  - Wisconsin Institute for Neurologic and Sleep Disorders, Milwaukee, Wisconsin
- Canada (8):
  - Movement Disorders Clinic, Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - Saint Boniface Clinic, Winnipeg, Manitoba
  - London Health Science Center, London, Ontario
  - Parkinson's and Neurodegenerative Disorders Clinic, Ottawa, Ontario
  - Ottawa Hospital Civic Site, Ottawa, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Memory and Motor Skills Clinic, Québec, Quebec
  - University of Sherbrooke, Sherbrooke, Quebec
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - West Tallin Central Hopsital, Tallinn
- Latvia (2):
  - P.Stradina university hospital, Riga
  - Gailezers hospital, Riga
- Lithuania (5):
  - Kaunas Medical University Hospital, Kaunas
  - Siauliai Regional Hospital, Šiauliai
  - Vilnius University Emergency Hospital, Vilnius
  - Vilnius University Centre of Gerontology and Rehabilitation, Vilnius
  - Vilnius University Hospital Santariskiu klinikos, Vilnius
- Romania (7):
  - Psychiatry and Neurology Hospital, Neurology Department, Brasov
  - Colentina Clinical Hospital Bucharest, II Neurology Department, Bucharest
  - County Emergency Clinical Hospital Cluj-Napoca, I Neurology Clinic, Cluj-Napoca
  - CFR Clinical Hospital Constanta, Constanța
  - Clinical Rehabilitation Hospital Iasi, Neurology Department, Iași
  - County Clinical Emergency Hospital, Targu Mures, II Neurology Department,, Târgu Mureş
  - County Clinical Emergency Hospital Timisoara, Timișoara
- Ukraine (9):
  - Neurology department of Regional hospital named after Mechnikov, Dnipro
  - Department of Psychiatry and Medical Psychology of Donetsk National Medical University, Donetsk
  - Department of Neurological Diseases and Medical Genetic of Donetsk National Medical University, Donetsk
  - 1st neurology department of Central Clinical Hospital of Ukrzaliznytsya, Kharkiv
  - Institute of Gerontology Parkinson's Disease Center, Kiev
  - Neurology department of Lviv regional clinical hospital, Lviv
  - Neurology department of Medical Dental Academy based on Poltava regional hospital, Poltava
  - Neurology department of Vinnitsa Medical University, Vinnitsa
  - Neurology department, Zaporozhye State Medical University, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pahwa R, Lyons KE, Hauser RA, Fahn S, Jankovic J, Pourcher E, Hsu A, O'Connell M, Kell S, Gupta S; APEX-PD Investigators. Randomized trial of IPX066, carbidopa/levodopa extended release, in early Parkinson's disease. Parkinsonism Relat Disord. 2014 Feb;20(2):142-8. doi: 10.1016/j.parkreldis.2013.08.017. Epub 2013 Sep 5. PMID 24055014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 4/13/2009 Last patient out 10/05/2010
Pre-assignment Details: Following enrollment, subjects were randomized into one of the four treatment groups.
Groups:
- Placebo: Placebo capsules were used
- IPX066 145 mg LD: IPX066 capsule containing 145 mg levodopa and 36.25 mg carbidopa
- IPX066 245 mg LD: IPX066 capsules containing 245 mg levodopa and 61.25 mg carbidopa
- IPX066 390 mg LD: IPX066 capsules that contained 390 mg levodopa and 97.5 mg carbidopa
Period: Overall Study
Arm/Group | Placebo | IPX066 145 mg LD | IPX066 245 mg LD | IPX066 390 mg LD
Started (Baseline) | 92 | 87 | 104 | 98
Week 4 | 88 | 79 | 94 | 86
Week 9 | 80 | 73 | 88 | 78
Week 16 | 74 | 73 | 87 | 74
Week 23 | 71 | 72 | 85 | 74
Completed (Week 30) | 71 | 72 | 83 | 74
Not Completed | 21 | 15 | 21 | 24
Not completed — Adverse Event | 4 | 5 | 15 | 15
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 12 | 4 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 4 | 3 | 1 | 3
Not completed — Noncompliance | 0 | 0 | 1 | 1
Not completed — Other | 1 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population is all treated
Groups:
- IPX066 145 mg LD: IPX066 capsules containing 145 mg levodopa and 36.25 mg carbidopa
- IPX066 390 mg LD: IPX066 capsules containing 390 mg levodopa and 97.5 mg carbidopa
- Total: Total of all reporting groups
Arm/Group | Placebo | IPX066 145 mg LD | IPX066 245 mg LD | IPX066 390 mg LD | Total
Number analyzed (Participants) | 92 | 87 | 104 | 98 | 381
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (9.43) | 63.8 (9.81) | 65.2 (9.73) | 64.8 (9.32) | 64.8 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 45 | 44 | 169
  Male | 52 | 47 | 59 | 54 | 212
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 7 | 4 | 19
  Not Hispanic or Latino | 87 | 78 | 91 | 89 | 345
  Unknown or Not Reported | 2 | 4 | 6 | 5 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 0 | 1 | 2
  Black or African American | 0 | 0 | 2 | 0 | 2
  White | 90 | 87 | 102 | 96 | 375
  Other | 1 | 0 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 9 | 9 | 9 | 37
  Latvia | 1 | 1 | 0 | 0 | 2
  Romania | 13 | 13 | 15 | 14 | 55
  United States | 30 | 29 | 37 | 38 | 134
  Ukraine | 28 | 29 | 32 | 26 | 115
  Lithuania | 7 | 4 | 8 | 8 | 27
  Estonia | 3 | 2 | 3 | 3 | 11
Age at Parkinson's disease onset [Mean (Standard Deviation); unit: years] | 63.7 (9.48) | 61.7 (10.71) | 63.6 (10.43) | 63.0 (9.38) | 63.0 (10.00)
Duration of Parkinson's disease [Mean (Standard Deviation); unit: years] | 1.8 (2.01) | 2.3 (3.08) | 1.8 (1.85) | 2.0 (2.33) | 2.0 (2.34)
UPDRS Parts II and III Score [Mean (Standard Deviation); unit: units on a scale] — Unified Parkinson's Disease Rating Scale (UPDRS) - Four Parts Higher score values represent a worse outcome.
  Subscales II and III were summed:
  Part I: Mentation, Behavior and Mood - 4 questions 1-4 Score range: 1-16 Part II: Activities of Daily Living - 13 questions 5-17 Score range: 0-52 Part III: Motor Examination - 19 questions 18-31 and 25 total assessments Score range: 0-100 Part IV: Complications of Therapy (In the past week) - 11 questions Score range: 0-25
  units on a scale | 36.3 (11.89) | 36.1 (13.56) | 38.1 (15.63) | 36.3 (13.04) | 36.7 (13.63)
Hoehn and Yahr Stage [Number; unit: units on a scale] — Hoehn and Yahr Staging of Parkinson's Disease: Stages move from 1 - 5 with the worse outcome stage being Stage 5.
  Stage 1 = Symptoms on one side of the body only. Stage 2 = Symptoms on both sides of the body, No impairment of balance. Stage 3 = Balance impairment. Mild to moderate disease. Physically independent. Stage 4 = Severe disability but still able to walk or stand unassisted. Stage 5 = Wheelchair bound or bedridden unless assisted.
  units on a scale
    Stage I | 7 | 6 | 13 | 14 | 40
    Stage II | 69 | 62 | 65 | 62 | 258
    Remaining | 16 | 19 | 26 | 22 | 83
MMSE [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Examination (MMSE) is a 30-point questionnaire that is used extensively to measure cognitive impairment. Any score greater than or equal to 24 points (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
  units on a scale | 28.9 (1.18) | 29.0 (1.27) | 28.7 (1.21) | 28.9 (1.18) | 28.9 (1.21)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Sum of UPDRS Part II + UPDRS Part III at Week 30
Description: Analysis of the Change from Baseline in the sum of the Unified Parkinson's Disease Rating Scale (UPDRS) Part II (Activities of Daily Living) + UPDRS Part III (Motor Examination) at Week 30 (End of Study).
  Unified Parkinson's Disease Rating Scale (UPDRS) - Four Parts Higher score values represent a worse outcome.
  Subscales II and III were summed:
  Part I: Mentation, Behavior and Mood - 4 questions 1-4 Score range: 1-16 Part II: Activities of Daily Living - 13 questions 5-17 Score range: 0-52 Part III: Motor Examination - 19 questions 18-31 and 25 total assessments Score range: 0-100 Part IV: Complications of Therapy (In the past week) - 11 questions Score range: 0-25
Time Frame: Week 30
Population: Analysis included all treated subjects with at least one efficacy measurement after dosing. Subjects who had no post-baseline efficacy assessments (N4) and those who had early termination assessments>3 days after last dose and no other post-baseline measurements (N16) were not included in the efficacy analysis set. Randomized (381)-(4+16) = 361.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IPX066 145mg LD: IPX066 capsules containing 145 mg levodopa and 36.25 mg carbidopa
Arm/Group | Placebo | IPX066 145mg LD | IPX066 245 mg LD | IPX066 390 mg LD
Number analyzed (Participants) | 90 | 82 | 99 | 90
units on a scale | -0.6 (10.37) | -11.7 (10.97) | -12.9 (11.42) | -14.9 (11.85)

2. Secondary Outcome: Summary of Change From Baseline to End of Study in Mean Parkinson's Disease Questionnaire-39 (PDQ-39) Score
Description: Change from Baseline in Parkinson's disease Questionnaire 39 (PDQ-39) at Weeks 4, 9, 16, 23 and 30 or early discontinuation was collected. The PDQ-39 is a self-reported questionnaire consisting of 39 questions regarding the subjects mobility and the responses consist of "Never" (better in outcome), (value 0), "Occasionally" (value 1), "Sometimes" (value 2), , "Often" (value 3), and "Always" (value 4), (worse in outcome). The minimum possible score is "0" and the maximum is "156". The outcome measure calculated was the change from baseline to end of study in mean PDQ-39 score. Negative values indicate a better result.
Time Frame: Baseline and Week 30 (or End of Study)
Population: Subjects who had no postbaseline efficacy assessments (N=4) and those who had early termination assessments >3 days after last dose and no other postbaseline measurements (N=16) were not included in the efficacy analysis. 2 subjects without a baseline measurement, 1 each from 145mg and 390mg arm were also excluded. Randomized 381-4-16-2=359.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPX066 145 mg LD | IPX066 245 mg LD | IPX066 390 mg LD | Placebo
Number analyzed (Participants) | 81 | 99 | 89 | 90
score on a scale | -4.4 (12.18) | -3.8 (12.16) | -6.0 (12.30) | 0.6 (11.10)

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Arm/Group | Placebo | IPX066 145 mg LD | IPX066 245 mg LD | IPX066 390 mg LD
Serious Adverse Events (participants affected / at risk) | 3/92 | 4/87 | 5/104 | 2/98
Other Adverse Events (participants affected / at risk) | 26/92 | 27/87 | 47/104 | 48/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=92) | IPX066 145 mg LD (N=87) | IPX066 245 mg LD (N=104) | IPX066 390 mg LD (N=98)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary Artery Bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=92) | IPX066 145 mg LD (N=87) | IPX066 245 mg LD (N=104) | IPX066 390 mg LD (N=98)
Nausea (Gastrointestinal disorders) | 8 | 12 | 20 | 20
Headache (Nervous system disorders) | 10 | 6 | 13 | 17
Dizziness (Nervous system disorders) | 5 | 8 | 20 | 12
Insomnia (Psychiatric disorders) | 3 | 2 | 9 | 6
Abnormal dreams (Psychiatric disorders) | 0 | 2 | 6 | 5
Dry Mouth (Gastrointestinal disorders) | 1 | 3 | 2 | 7
Vomiting (Gastrointestinal disorders) | 3 | 2 | 2 | 5
Constipation (Gastrointestinal disorders) | 1 | 2 | 6 | 2
Dyskinesia (Nervous system disorders) | 0 | 2 | 4 | 5
Anxiety (Psychiatric disorders) | 0 | 2 | 3 | 5
Depression (Psychiatric disorders) | 5 | 1 | 2 | 2
Orthostatic Hypotension (Vascular disorders) | 1 | 1 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results of the Study conducted at the Site shall not be made before the first multi-site publication by Sponsor.